CLINICAL TRIAL: NCT00001428
Title: A Phase II Study of 5-Fluorouracil Administered as a One Hour Infusion in Combination With Calcium Leucovorin and Interferon Alpha-2A in Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950067; 95-C-0067
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Colorectal Neoplasms
Keywords: Chemotherapy; Cytokine; Efficacy; Palliation; Solid Tumor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil

INTERVENTIONS:
Drug: 5-fluorouracil

SUMMARY:
This protocol will evaluate the activity of 5-Fluorouracil (FUra) given as a 1 hour infusion in combination with leucovorin (LV) and interferon IFN alpha-2a in patients with advanced, measurable colorectal cancer.

DETAILED DESCRIPTION:
This protocol will evaluate the activity of 5-Fluorouracil (FUra) given as a 1 hour infusion in combination with leucovorin (LV) and interferon IFN alpha-2a in patients with advanced, measurable colorectal cancer. IFN alpha-2a will be given at 5 million U/m(2) SC days 1-6; LV, 200 mg/m(2), will be given as a short infusion over 30 minutes days 2-6, followed immediately by a 1 hour IV infusion of FUra days 2-6. The starting dose of FUra will be 425 mg/m(2)/d(1). Cycles will be repeated at three week intervals provided that the granulocyte count and platelet count have recovered to &gte; 1200/microL and &gte; 80,000/microL, respectively, and all non-hematologic toxicity has resolved. The dose of FUra will be adjusted according to individual tolerance. Preliminary experience with FUra given as a 1 hour infusion suggests that it is less toxic. The primary goal of this study is to determine if this less toxic regimen retains clinical antitumor activity. FUra plasma samples will be obtained the initial cycle at 50 and 55 minutes during the first 1 hour infusion of FUra to permit documentation of achieved plasma levels and to permit correlation between FUra pharmacokinetics and clinical toxicity and/or response. Pharmacokinetic sampling will be repeated if the dose of FUra is increased or decreased in subsequent cycles.

Patients will be stratified according to whether or not they have received prior adjuvant chemotherapy. A two-stage design will be employed for patients with no prior chemotherapy: If less than or equal to 4 responses are seen among the initial 20 previously untreated patients, accrual will cease. If greater than or equal to 5 responses are seen in the initial 20 patients, however, accrual will be expanded to 40 patients.

Fourteen patients who have received prior adjuvant chemotherapy (completing it at least 6 months prior to study entry) or have received prior FUra only as a radiation sensitizer will be entered. If no responses are seen, accrual to this cohort will cease. If greater than or equal to 1 response is seen, accrual may be expanded to 24 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Unresectable primary colorectal adenocarcinoma that is metastatic or recurrent.

Objectively measurable disease required.

No cerebral metastases.

PRIOR/CONCURRENT THERAPY:

Biologic Therapy:

No history of intolerance to interferon alfa (IFN-A).

At least 4 weeks since immunotherapy and recovered.

Chemotherapy: No prior chemotherapy for metastatic or recurrent disease. At least 6 months since adjuvant chemotherapy with fluorouracil (5-FU) in combination with levamisole, leucovorin (CF), or IFN-A Interval waived for 5-FU (with or without CF) as a radiosensitizer only . No dose-limiting toxicity with prior 5-FU.

Endocrine Therapy: Not specified

Radiotherapy: At least 2 weeks since palliative radiotherapy and recovered. Prior definitive pelvic or whole or upper abdominal radiotherapy allowed in the absence of current radiation enteritis.

Surgery: Prior surgery allowed with adequate healing/recovery

Patient Characteristics:

Age: 18 and over.

Performance status: ECOG 0 or 1.

Hematopoietic:

AGC at least 2,000.

Platelets at least 100,000.

Hepatic: Bilirubin no greater than 2.0 mg/dL

Renal: Creatinine no greater than 2.0 mg/dL

Cardiovascular:

No MI within the past year.

No active ischemic heart disease.

No NYHA class III/IV status.

No symptomatic arrhythmia.

OTHER:

No requirement for pharmacologic steroid doses for inflammatory or autoimmune disorders. Physiologic replacement doses of steroids allowed.

No concurrent cimetidine or oxypurinol.

No HIV antibody.

No history of seizure disorder.

No active infection or other serious concurrent medical illness that would preclude treatment.

No second malignancy within 3 years except curatively treated: In situ carcinoma of cervix, Basal cell carcinoma of the skin.

No pregnant or nursing women.

Effective contraception required of fertile patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 1995-02; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Miyoshi T, Ogawa S, Kanamori T, Nobuhara M, Namba M. Interferon potentiates cytotoxic effects of 5-fluorouracil on cell proliferation of established human cell lines originating from neoplastic tissues. Cancer Lett. 1983 Jan;17(3):239-47. doi: 10.1016/0304-3835(83)90160-x. PMID 6187435
- [Background] Le J, Yip YK, Vilcek J. Cytolytic activity of interferon-gamma and its synergism with 5-fluorouracil. Int J Cancer. 1984 Oct 15;34(4):495-500. doi: 10.1002/ijc.2910340411. PMID 6436183
- [Background] Elias L, Crissman HA. Interferon effects upon the adenocarcinoma 38 and HL-60 cell lines: antiproliferative responses and synergistic interactions with halogenated pyrimidine antimetabolites. Cancer Res. 1988 Sep 1;48(17):4868-73. PMID 2457431